CLINICAL TRIAL: NCT06938737
Title: Effects of Laughter Yoga on Happiness, Mental Well-being and Blood Pressure in Hemodialysis Patients: A Randomized Controlled Trial
Brief Title: Laughter Yoga Intervention in Patients on Haemodialysis
Acronym: laughter yoga
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Füsun UZGÖR, dr research assistant, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 240045
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Haemodialysis Patients; Laughter Yoga
Keywords: Haemodialysis; laughter yoga; Happiness; Mental Well-being; blood pressure
MeSH Terms: conditions — Psychological Well-Being | interventions — Laughter Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): Both groups of patients will complete the Introductory Information Form, Blood Pressure Monitoring Form, Oxford Happiness Scale and Warwick-Edinburgh Mental Well-Being Scale for the first assessment.
  In addition to routine treatment and care, patients in the application group will receive a total of 8 sessions of laughter yoga, each session lasting approximately 30 minutes, once a week for 8 weeks by a researcher with a directed self-determination method certificate.
  The patients' blood pressure will be monitored and recorded before and after each laughter yoga session.
  Blood pressure monitoring form, Oxford Happiness Scale and Warwick-Edinburgh Mental Well-being Scale will be applied to the patients in the 4th week and 8th week.
  Interventions: Behavioral: laughter yoga
- Control group (No Intervention): Both groups of patients will complete the Introductory Information Form, Blood Pressure Monitoring Form, Oxford Happiness Scale and Warwick-Edinburgh Mental Well-Being Scale for the first assessment.
  Patients will receive routine treatment and care. Blood pressure monitoring form, Oxford Happiness Scale and Warwick-Edinburgh Mental Well-being Scale will be applied to the patients in the 4th week and 8th week.

INTERVENTIONS:
Behavioral: laughter yoga — Laughter yoga sessions begin with gentle warm-up techniques that include stretching and flexing movements, songs, applause and body movements. These techniques aim to break down any inhibitions against laughter and develop childlike playfulness. Breathing exercises prepare the lungs for laughter and are combined with a series of laughter exercises that follow.
  Arms: intervention group

SUMMARY:
This study was planned as a randomized controlled experimental type and pre-test-post-test design in order to examine the effects of laughter yoga applied to hemodialysis patients on the happiness and mental well-being levels of the patients and on blood pressure.

The universe of the study will be patients receiving hemodialysis treatment at Fethiye Özel Can Dialysis Center (N=184) and the sample will be a total of 72 patients, consisting of the experimental group (n=36) and the control group (n=36).

After obtaining the permission of the ethics committee and institution, the data will be collected face to face by the researchers before and after the laughter yoga to be applied to hemodialysis patients receiving treatment at Fethiye Özel Can Dialysis Center and who agreed to participate in the study. In the collection of data; Introductory Information Form (TBF), Warwick-Edinburgh Mentai Well-Being Scale (WEMİOÖ), Oxford Happiness Scale (OMÖ) and blood pressure measurements of the patients will be used. IBM SPSS 25.0 package program will be used to evaluate the data.

DETAILED DESCRIPTION:
Chronic renal failure (CRF) is defined as a permanent decrease in glomerular filtration rate due to progressive deterioration of renal functions as a result of progressive nephron loss in the patient or as a damage condition accompanied by structural or functional disorders lasting longer than three months in the kidneys regardless of glomerular filtration. The renal replacement therapy method commonly used in the treatment of chronic renal failure is hemodialysis. Although hemodialysis increases the life expectancy of patients, with the inclusion of hemodialysis in patients' lives; their mental state, family relationships, work life, social relationships and roles are affected, and a decrease in their emotional performance is experienced. As a result of being dependent on the dialysis device, family and healthcare team during the treatment process, which has become an important part of patients' lives; sadness, anger, hopelessness, anxiety, helplessness, fluid restriction, pain, cramps, nausea, limited diet, introversion, decreased self-confidence, anxiety about becoming dependent, depression, body image changes, social isolation, sleep disorders, sexual dysfunction, lifestyle deterioration, fear of the future and death, and many other physical and psychosocial problems are experienced. Happiness is one of the determinants of mental health, which plays an important role in shaping a person's personality and mental health. Happiness, defined as a series of emotions and cognitive evaluations of life, is accepted as a degree that shows that the quality of life is positive. Mental well-being is defined as "the individual being aware of his/her own abilities, being able to overcome the stress in his/her life, being productive and useful in his/her life and contributing to the society in line with his/her abilities". Studies have shown that individuals with high levels of mental well-being have better psychological and physical health and higher quality of life.

Blood pressure changes frequently seen in patients receiving hemodialysis treatment negatively affect the lives of individuals. In particular, the increased symptom load due to intradialytic hypotension negatively affects the quality of life of patients.

Laughter yoga is a non-invasive and non-pharmacological therapy method that combines unconditional laughter with breathing techniques. It has been reported that laughter yoga physiologically in the body; increases breathing, relaxes muscles, stimulates circulation and the immune system, improves vascular endothelial function, regulates blood pressure, increases pain threshold and pain tolerance by increasing endorphin hormone release, strengthens mental functions by reducing the level of stress hormones; reduces depression and anxiety levels, improves sleep quality, and provides psychological well-being by increasing interpersonal relationships and social interaction.

This study was planned as a randomized controlled experimental type and pre-test-post-test design in order to examine the effects of laughter yoga applied to hemodialysis patients on the happiness and mental well-being levels of the patients and on blood pressure.

The universe of the study will be patients receiving hemodialysis treatment at Fethiye Özel Can Dialysis Center (N=184) and the sample will be a total of 72 patients, consisting of the experimental group (n=36) and the control group (n=36).

After obtaining the permission of the ethics committee and institution, the data will be collected face to face by the researchers before and after the laughter yoga to be applied to hemodialysis patients receiving treatment at Fethiye Özel Can Dialysis Center and who agreed to participate in the study. In the collection of data; Introductory Information Form (TBF), Warwick-Edinburgh Mentai Well-Being Scale (WEMİOÖ), Oxford Happiness Scale (OMÖ) and blood pressure measurements of the patients will be used. IBM SPSS 25.0 package program will be used to evaluate the data.

ELIGIBILITY:
Inclusion Criteria:

1. Those receiving hemodialysis treatment at Fethiye Can Dialysis Center with a diagnosis of CKD
2. 18 years of age and older
3. Ability to read and understand
4. Those receiving hemodialysis treatment for six months or longer
5. Interdialytic fluid intake not more than 5% of total weight
6. Able to communicate in Turkish
7. No hearing or vision loss
8. Patients who volunteer to participate in the study

Exclusion Criteria:

1. Those with interdialytic fluid intake greater than 5% of total weight
2. Those with respiratory system diseases that negatively affect the practice of laughter yoga (COPD, asthma, bronchiectasis, lung infections, etc.)
3. Those with hearing and vision loss
4. Those who want to leave the study despite completing the survey questions appropriately
5. Those who do not agree to participate in the study
6. Those aged 18 and under
7. Those who start treatment at another dialysis center
8. Those who change their renal replacement therapy type -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-04-28 (Estimated); Primary Completion 2025-06-16 (Estimated); Study Completion 2025-06-20 (Estimated)

PRIMARY OUTCOMES:
The change in happiness levels in patients on haemodialysis | week 0, week 4, week 8
  Happiness will be evaluate in study with the Oxford Happiness Questionnaire. This scale consists of 29 questions and is a six-point Likert type question "I do not agree at all, I mostly disagree, I somewhat agree, I agree, I mostly agree and I completely agree". The lowest score that can be obtained from the scale is 29 and the highest score is 145. In addition, as the score obtained from the scale increases, the level of happiness also increases. The Cronbach Alpha value of the scale was obtained as 0.91
The change in mental well-being level in patients on haemodialysis | week 0, week 4, week 8
  The mental well-being level will be evaluated with the Warwick-Edinburgh Mental Well-Being Scale. The scale is a 5-point Likert type and the minimum score is 14 and the maximum score is 70. High scores obtained from the scale indicate high mental (psychological) well-being. The scoring of the scale is (1=I do not agree at all, 2=I do not agree, 3=I somewhat agree, 4=I agree, 5=I completely agree). All items of the scale are positive. The Cronbach alpha internal consistency reliability coefficient of the scale was found to be .92.
blood pressure | 16 times in total before and after each session (twice a week for 8 weeks)
  Blood pressure of patients will be monitored before and after laughter yoga and recorded on the blood pressure monitoring form.

CONTACTS AND LOCATIONS:
Locations (1):
- Mugla Sıtkı kocman University, Muğla, Turkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1- Akpınar NB, Ceran BA. (2019). Kronik Hastalıklar ve Rehabilitasyon Hemşireliği. Adnan Menderes Üniversitesi Sağlık Bilimleri Fakültesi Dergisi. 3(2): 140-152. 2- Akpınar NB, Ceran MA, Şafak Ş, Özkalp B. (2019). Hemodiyaliz hastalarının öz yeterlilik durumu, bakım gereksinimi ve günlük yaşam aktivitelerini gerçekleştirebilme düzeyleri. Hemşirelik Bilimi Dergisi, 2 (1): 5-10. 3- Becerra LC, Garcia-Molina M. (2015).Happiness Effects on Health-State Valuations. Value in Health, 18(7):A716. 4- Bennett PN, Parsons T, Ben-Moshe R, Neal M, Weinberg MK, Gilbert K, Ockerby C, Rawson H, Herbu C, Hutchinson AM. (2015). Intradialytic Laughter Yoga therapy for haemodialysis patients: a pre-post intervention feasibility study. BMC Complement Altern Med. 9;15:176. doi: 10.1186/s12906-015-0705-5. 5- Bennett P.N., Weinberg M.K., Bridgman T., Cummins R.A. (2015). The happiness and subjective well-being of people on haemodialysis. Journal of Renal Care 41(3), 156-161. 6- Billington E, Simpson J, Unwin J, Bray D, Giles D.(2008). Does hope predict adjustment to end-stage renal failure and consequent dialysis? British journal of health psychology, 13(4):683-99. 7- Demiroğlu S, Bülbül E. (2021). Hemodiyaliz tedavisi alan hastaların depresyon, anksiyete, stres durumları ve diyaliz semptomlarıyla ilişkisi. Nefroloji Hemşireliği Dergisi, 16 (3): 124-133 8- Doğan, T., Sapmaz, F. (2012). Oxford mutluluk ölçeği türkçe formunun psikometrik özelliklerinin üniversite öğrencilerinde incelenmesi. Düşünen Adam Psikiyatri ve Nörolojik Bilimler Dergisi. 25(4), 297-304.https://doi.org/10.5350/DAJPN201225040. 9- El Filali A, Bentata Y, Ada N, Oneib B. (2017). Depression and anxiety disorders in chronic hemodialysis patients and their quality of life: A cross-sectional study about 106 cases in the northeast of morocco. Saudi Journal of Kidney Diseases and Transplantation, 28 (2): 341-348. 10- Fard Tabatabaei M, Raghibi M. (2017). Effect of happiness training in depression, anxiety, and quality of li